CLINICAL TRIAL: NCT00415402
Title: Randomised Controlled Trial to Evaluate the Preventive Effect on Mortality and Serious Morbidity/ Hospitalisations of Daily Vitamin D Supplements in Small for Gestational Age Term Infants
Brief Title: Effect of Vitamin D Supplementation on Health of Low Birth Weight Infants
Acronym: DIVIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delhi University (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Sitaram Bhartia Institute of Science and Research (Other)
Responsible Party: Principal Investigator, Dr Geeta Trilok-Kumar, Associate professor, Delhi University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BT/PR 7489/PID/20/285/2006; IHE/VITD/2006
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D3; morbidity; mortality; low birth weight; supplementation; TH1; TH2; CRP; Neopterin; immune response
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): non vitamin D containing sugar granules
- Vitamin D3 (Experimental): vitamin D granules
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3
  Arms: Vitamin D3

SUMMARY:
The purpose of this study is to determine whether a weekly supplement of vitamin D to low birth weight term infants will reduce their mortality and hospital admissions and improve their immunity.

DETAILED DESCRIPTION:
We are conducting a randomised controlled trial of weekly oral vitamin D supplements to low birth weight (< 2.5 kg) term infants born in a large government hospital catering to a low-middle income population in Delhi. Mothers and infants are recruited at delivery and given weekly vitamin D supplements or placebo until 6 months of age. Data on infant morbidity, sun exposure and diet, with particular emphasis on breast milk and other milk intake, is collected by fieldworkers visiting the homes each fortnight. Mothers are encouraged to bring their infants to the hospital in case of any illness and at these visits the infant is seen by the project doctor who treats the infant and records additional morbidity data. At 6 months blood samples are being collected from a 20% random subsample of infants for measurement of 25OHD and indicators of immune activation. The primary outcome is mortality or incidence of any illness requiring admission to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Born at term, as determined from last menstrual period
* Weighing < 2.5 kg
* Resident within 12 km of the hospital and expected to continue living in the area for the following 6 months
* With no severe congenital abnormalities
* No morbidity severe enough to be expected to result in death before 7 days due to severe respiratory distress, shock, pulmonary sepsis, etc.
* Parental informed consent

Ages: 24 Hours to 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Actual)
Dates: Start 2007-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Mortality | weekly
Incidence of disease requiring hospitalization
Morbidity and hospitalization | weekly

SECONDARY OUTCOMES:
Incidence of infectious disease not requiring hospitalization
Severe morbidity requiring hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Geeta Trilok-Kumar, PhD, Principal Investigator — Institute of Home Economics, Delhi University
Locations (1):
- Institute of Home Economics, Delhi University, New Delhi, India

REFERENCES:
- [Result] Kumar GT, Sachdev HS, Chellani H, Rehman AM, Singh V, Arora H, Filteau S. Effect of weekly vitamin D supplements on mortality, morbidity, and growth of low birthweight term infants in India up to age 6 months: randomised controlled trial. BMJ. 2011 May 31;342:d2975. doi: 10.1136/bmj.d2975. PMID 21628364
- [Result] Trilok-Kumar G, Arora H, Rajput M, Chellani H, Singh V, Raynes J, Arya S, Aggarwal S, Srivastava N, Sachdev HP, Filteau S. Effect of vitamin D supplementation of low birth weight term Indian infants from birth on cytokine production at 6 months. Eur J Clin Nutr. 2012 Jun;66(6):746-50. doi: 10.1038/ejcn.2012.33. Epub 2012 Apr 18. PMID 22510791
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842